CLINICAL TRIAL: NCT02749500
Title: Early Independent Adaptive Arm and Hand Rehabilitation Post Stroke
Brief Title: Early Independent Adaptive Arm and Hand Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-01460
Record Dates: First submitted 2016-04-15; First posted 2016-04-25 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Post-stroke Hemiparesis
Keywords: Motor control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Occupational Therapy (OT) (Active Comparator): Standard of care occupational therapy for stroke recovery
  Interventions: Other: Conventional Occupational Therapy (OT)
- OT + Device-assisted therapy (Experimental): Conventional OT plus 1 hour additional bimanual-to-unimanual device-assisted therapy. The m2 BAT will enable repeated movement of the affected body part without the help of a therapist, providing the opportunity to maintain range-of motion in the affected limb to limit spasticity, contracture and the ensuing deformity, a major goal of rehabilitation therapy and produces movement in the affected limb from activating the patient's own brain, rather than from being acted on by an external powered source such as a robot.
  Interventions: Other: Conventional Occupational Therapy (OT); Device: m2 BAT

INTERVENTIONS:
Other: Conventional Occupational Therapy (OT) — Standard of care occupational therapy for stroke recovery
Device: m2 BAT — Conventional OT plus 1 hour additional bimanual-to-unimanual device-assisted therapy.
  Arms: OT + Device-assisted therapy

SUMMARY:
The purpose of this study is to test the hypothesis that early independent adaptive bimanual-to-unimanual training of arm and hand movements, assisted with specially designed mechanical devices: the mirrored motion bimanual arm trainer (m2 BAT), will improve motor control and function in patients with post-stroke hemiparesis.

DETAILED DESCRIPTION:
This study will randomly assign individuals admitted to the inpatient stroke rehabilitation unit to receive either conventional occupational therapy (OT) or conventional OT plus 1 hour additional bimanual-to-unimanual device-assisted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to follow study instructions
* Ability to likely complete all required visits
* Ability to comply with the therapy protocol as assessed by the investigator
* Must be English speaking
* Subjects must have had a unilateral stroke

Exclusion Criteria:

* Severe upper extremity spasticity suggested by an Ashworth score of ≥3 at any joint, or restriction of full passive range of motion.
* Evidence of alcohol, drug abuse or other relevant neuropsychiatric condition such as psychotic illness or severe depression.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* History of surgery or other significant injury to either upper extremity causing mechanical limitations that preclude task performance.
* Previous neurological illness such as head trauma, prior stroke, epilepsy, or demyelinating disease.
* Complicating medical problems such as uncontrolled hypertension, diabetes with signs of polyneuropathy, severe renal, cardiac or pulmonary disease, or evidence of other concurrent neurologic or orthopedic conditions precluding the subject from complying with the study protocol.
* Patients who are cognitively impaired.
* Patients who lack capacity to consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
Performance tasks of the Fugl-Meyer Scale (FMS) | 12 Weeks
  This measurement will be on a 3-point ordinal scale, ranging from 0-2 with a maximum score of 66.
Upper extremity functional ability measured with Modified Rankin Scale | 12 Weeks
Stroke-related quality of life measured with the Stroke Impact Scale | 12 Weeks
Spasticity measured using the Modified Ashworth Scale | 12 Weeks
Range of motion will be measured using video | 12 Weeks
  Active/passive range of motion for shoulder flexion, extension, abduction, internal and external rotation, elbow flexion and extension, pronation and supination, wrist flexion and extension, radial and ulnar deviation will be measured for affected and unaffected arms.
Upper extremity functional ability measured using the Wolf Motor Function Test | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Tafurt, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States